CLINICAL TRIAL: NCT07139925
Title: Validation of a Self-Care Assessment Tool for Patients With Idiopathic Pulmonary Fibrosi
Brief Title: Assessment of Self-Care in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: SC-IPFI
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RICHELDI LUCA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7153
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: IPF

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self-care of COPD Inventory (SC-COPDI) — Self-care of COPD Inventory (SC-COPDI) - Assess the self-care of patients with IPF by adapting a tool designed for patients with COPD to those affected by IPF

SUMMARY:
The adaptation of the SC-COPDI for IPF patients

DETAILED DESCRIPTION:
Cross-sectional, single-center observational study. The study aims to adapt a tool designed for patients with COPD (SC-COPDI) for use with patients affected by idiopathic pulmonary fibrosis

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic pulmonary fibrosis (IPF)
* Patients over 18 years of age
* Patients who are able to provide informed consent to participate in the study

Exclusion Criteria:

* Patients diagnosed with cognitive impairment
* Patients who are unable to speak, read, or write in Italian
* Patients who are blind or deaf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with idiopathic pulmonary fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of a tool for assessing self-care in patients with IPF | baseline
  To make a tool available for assessing self-care in patients with IPF by adapting an instrument designed for patients with COPD to those with IPF

CONTACTS AND LOCATIONS:
Overall Officials: Luca Richeldi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Roma, Roma, Italy